CLINICAL TRIAL: NCT07182747
Title: Feasibility of a Multidisciplinary Intervention Programme Carried Out by Nursing and Physical Activity and Sports Sciences Students to Improve Frailty and Other Related Variables in Older Adults Living in Nursing Homes.
Brief Title: Feasibility of a Multidisciplinary Student-Led Program to Improve Frailty in Nursing Home Residents
Acronym: CUIDAFRAIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Jose Manuel Hernandez Padilla, Professor (Full), Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01037772
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Frailty
Keywords: Frailty; older adults; intervention programme; Physical Activity; Activities of Daily Living; Nursing student; feasibility
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Older adults who meet the inclusion criteria and voluntarily accept to participate in this study will be randomly allocated to one of two arms: intervention group (arm 1) or control group (arm 2). Participants from both arms will be assessed at the same time for data collection purposes (pre-test, post-test and 6-month follow-up) and they will be exposed to the experimental condition (intervention group) or the control condition (control group) at the same time for 12-weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The type of intervention on which the project is based does not allow for the participants to be masked and they will know to which group they are allocated. However, the team that will collect data (assessors) will not know the group to which each participant is allocated. To ensure assessor masking, participants will be instructed to never reveal the group to which they have been assigned and assessors will be instructed to never ask the participants to which group they have been assigned. The assessors will not participate in the recruitment process, the supervision of nursing students' interventions, nor the data analysis process. The group to which the participants have been allocated will be numerically coded (not labelled) in the database and the researchers in charge of data analysis will not know which numerical code refers to the intervention group and which code refers to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants allocated to the 'intervention group' arm will receive the usual care offered by the Public Andalusian Healthcare Service in conjunction with a 12-week nursing students' intervention programme.
  Interventions: Behavioral: Nursing students' intervention programme; Behavioral: Standard care from Public Andalusian Health Service
- Control group (Active Comparator): Participants allocated to the 'control group' arm will only receive the usual care offered by the Public Andalusian Healthcare Service for 12 weeks.
  Interventions: Behavioral: Standard care from Public Andalusian Health Service

INTERVENTIONS:
Behavioral: Nursing students' intervention programme — 12-week intervention programme conducted by nursing students and students trained in Sciences of Physical Activity and Sport (CAFYD). Participants will receive weekly three sessions of 45-60 minutes. It will include physical exercise and occupational therapy sessions aimed at improving frailty and other related outcomes in the participating older adults through interdisciplinary collaboration and ongoing monitoring. Nursing students will implement personalised intervention programmes designed by a multidisciplinary team comprising CAFYD students, an occupational therapist, and nurses experienced in the care of older adults.
  Arms: Intervention group
Behavioral: Standard care from Public Andalusian Health Service — They will receive the standard care provided by the Andalusian Health Service as part of its portfolio of services offered to older adults residing in institutions, as well as the standard care provided by the institutions in which they live. As part of these services, older adults receive support such as accommodation, laundry, health promotion activities, health monitoring, assistance with activities of daily living, individual, group, and community social care, as well as means of communication with the outside world. The action plans or protocols established in care processes for older adults living in nursing homes do not include externally delivered multidisciplinary intervention programmes.

SUMMARY:
BACKGROUND Frailty, regarded as a potentially reversible process and defined as a progressive deterioration of physiological systems and intrinsic capacity, constitutes a key risk factor for disability, dependency and institutionalisation.

Currently, it is estimated that between 50% and 75% of older adults living in residential care facilities present with frailty. This clinical profile is often directly associated with multiple comorbidities (around 65-85% of this population suffer from several chronic conditions), emotional decline, polypharmacy, malnutrition and a high prevalence of functional and cognitive impairment. Consequently, two out of every three older adults will require long-term care in specialised centres during their lifetime. In this context, nursing homes represent a key setting not only for providing care, but also for the prevention, detection and management of conditions such as frailty. However, care in residential facilities continues to focus on addressing established problems, with low participation in activities with potential benefits and a high perception of loneliness. Therefore, interventions in these contexts aimed at improving frailty are both necessary and urgent, particularly those that integrate a biopsychosocial approach, promote autonomy and foster active ageing.

Several studies have demonstrated that multidisciplinary intervention programmes and multicomponent physical training are effective in preventing frailty and its consequences. Nevertheless, their widespread implementation is limited by several factors. On the one hand, there is a lack of scientific evidence on the cost-effectiveness of such interventions, and on the other, healthcare systems face budgetary constraints in a context of increasing demand for geriatric care. In the search for more effective interventions to improve frailty and other related variables in older adults residing in nursing homes, supervised multidisciplinary programmes, delivered by health sciences students and implemented by nursing students, may represent a viable alternative. In this regard, students of Physical Activity and Sport Sciences (CAFYD) possess the knowledge required to design physical activity plans adapted to the capacities and needs of older adults. However, given the nature of their care role, nurses provide added value: their continuous presence in the clinical setting enables them to establish a closer therapeutic bond with the patient, ensure thorough monitoring of their progress, and facilitate coordination between physicians and other healthcare team members. These features make nurses key agents in the implementation of comprehensive, person-centred interventions.

Despite the potential of implementing a multidisciplinary intervention programme through health sciences students to improve frailty in older adults living in residential facilities, to the best of our knowledge, no similar interventions exist. Therefore, it is necessary to assess the feasibility of implementing such a proposal prior to conducting a randomised controlled trial to confirm its clinical effectiveness, as this approach plays an important role in determining the most appropriate trial design. To this end, different feasibility study guidelines recommend including variables such as acceptance, adherence and dropout rates as key markers for successful implementation.

STUDY'S HYPOTHESIS The main hypothesis of the CUIDAFRAIL project is that a supervised multidisciplinary intervention programme carried out by nursing and Physical Activity and Sport Sciences students is feasible for improving frailty and other related variables in older adults living in residential care facilities.

AIM AND OBJECTIVES The aim of the CUIDAFRAIL project is to examine the short- term and medium-term effects of a nursing students' multidisciplinary intervention programme on frailty among older adults living in nursing homes.

The secondary objectives of this project are the following:

1. To examine the effects of the intervention on frailty, as well as other frailty-related variables, including physical fitness, functionality, fear of falling, emotional status, loneliness, social support and quality of life in older adults living in residential care facilities.
2. To examine the effects on physiological and clinical parameters associated with frailty.
3. To explore the perceptions and experiences of older adults participating in the programme upon completion.
4. To explore the perceptions and experiences of nursing and Physical Activity and Sport Sciences students upon completion of the programme.

STUDY DESIGN A feasibility study will be carried out. Participants will be randomly assigned to either an intervention group (IG) or a control group (CG).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Living in one of the institutions participating in the study.
* Signing the informed consent to participate in the study.

Exclusion Criteria:

* Requiring palliative care
* Having moderate or severe cognitive impairment (Pfeiffer Test >4); hypotension (systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg), anemia (hemoglobin level <9 g/dL), any acute metabolic disorder, uncontrolled hypertension (systolic blood pressure >160 mmHg, diastolic blood pressure >100 mmHg), uncontrolled arrhythmia, stable/unstable angina, uncontrolled chronic or metabolic disease, and advanced cerebrovascular or peripheral vascular disease
* Having undergone surgery within the last six weeks.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Adoption | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  The proportion of older adults who agree to participate out of the total number of older adults offered the programme. This information will be obtained from the records of eligible individuals and those ultimately included.
Adherence | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Adherence: The proportion of participants who complete at least 8 of the 12 weeks comprising the entire programme.
Dropout | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  The proportion of participants who withdraw from the intervention out of the total number of individuals who agreed to participate and began the programme.
Perceived quality of the intervention | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Assessed using the Net Promoter Scale (NPS), a tool used to measure user satisfaction with an intervention through the question: "How likely are you to recommend this to someone in a similar situation?" Scores range from 0 to 10, with scores below 5 indicating dissatisfaction and scores above 5 indicating satisfaction.
Frailty | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Clinical Frailty Scale (CFS). The CFS is a clinician-administered scale comprising nine levels that classify patients' degree of frailty. Each level describes a set of characteristics related to physical condition, functionality, and cognitive status, ranging from 1 (very fit) to 9 (terminally ill). Scores are assigned based on the patient's overall functioning in daily life, including mobility, dependence for basic and instrumental activities of daily living, presence of chronic diseases, and cognitive impairment. The scale has been validated in residential settings and can also be used in individuals with cognitive impairment, as it does not require self-reporting. Higher scores indicate greater frailty.

SECONDARY OUTCOMES:
Physical condition (SPPB total score) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be evaluated using the Short Physical Performance Battery (SPPB). The SPPB assesses the ability to maintain balance for 10 seconds in different positions, the time required to walk 4 metres, and the time required to rise from a chair five times. Each test is scored from 0 to 4, where 4 indicates the highest performance and 0 indicates an inability to complete the test. The total battery score ranges from 0 (worst performance) to 12 (best performance).
Physical condition (Timed Up and Go test) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Additionally, the Timed Up and Go (TUG) test will be used due to its association with fall risk. This test measures the time a participant takes to rise from a chair, walk 3 metres at their usual pace in a straight line, and return to a seated position. Shorter TUG times are considered indicative of better performance. A time exceeding 12 seconds is considered high fall risk; 10-12 seconds indicates moderate risk; and times below 10 seconds generally reflect good mobility and low fall risk.
Leg strength | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Leg strength will be assessed using the modified thirty-second chair stand test (m-30s-CST). Participants will be asked to sit in a chair with armrests of identical dimensions for all participants. They will attempt to rise from the chair to a full standing position as many times as possible within 30 seconds. Completing 10 or more repetitions indicates good leg strength and high mobility; 8-9 repetitions correspond to moderate strength and mobility; fewer than 8 repetitions indicate low leg strength and may be associated with increased fall risk.
Grip strength | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Grip strength will be evaluated given its documented correlation with frailty. It will be measured using a digital hand dynamometer (TAKEI TKK-5401) unilaterally, distinguishing between dominant and non-dominant hand.
Fall risk | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  The Downton Fall Risk Index will be used. This instrument comprises five sections assessing: previous falls, medication (particularly psychotropic drugs), sensory deficits, mental status, and gait. Each item has a specific score, and the total sum provides an estimate of overall fall risk. Each item can be scored 0 or 1, with a total score of 3 or more indicating a high risk of falls.
Functionality | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be measured using the Measure of Functional Independence (MIF). The scale includes 18 items, 13 of which are related to physical activities divided into four categories: self-care, continence, transfers, and mobility. The remaining five items assess cognitive and social aspects, divided into communication and social cognition categories. Total scores range from 18 to 126, with higher scores indicating greater independence. The psychometric properties of the MIF are adequate.
Fear of falling | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be assessed using the Short Falls Efficacy Scale-International (SFES-I), a quick and easy-to-administer scale with seven items related to different activities of daily living (ADLs) both inside and outside the home. Each item is scored from 1 (not at all concerned about falling during the activity) to 4 (very concerned about falling during the activity). Total scores range from 7 (no concern about falling) to 28 (extremely concerned).
Nutritional status | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Nutritional status will be assessed using the Short Form Mini Nutritional Assessment (MNA-SF). This consists of six brief questions covering key aspects of nutritional status. Total scores (maximum 14 points) classify participants as: normal nutritional status (12-14 points), at risk of malnutrition (8-11 points), or malnourished (0-7 points).
Cognitive status | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Cognitive function will be evaluated using the Mini-Mental State Examination (MMSE). This questionnaire assesses five dimensions: orientation, attention and calculation, memory, language, and praxis. Results are interpreted as follows: >24 points indicates no cognitive impairment, 19-23 points mild cognitive impairment, 14-18 points moderate cognitive impairment, and <14 points severe cognitive impairment.
Pain level | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Pain will be assessed using the Pain Assessment in Advanced Dementia (PAINAD) scale. This evaluates five items: breathing, negative vocalisation, facial expression, body language, and consolability. Scores correspond to: 0-4 points mild pain, 5-7 points moderate pain, and 8-10 points severe pain. This scale can be used in patients with or without cognitive impairment.
Prediction of pressure ulcer risk | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  The Braden Scale will be used. This scale evaluates six dimensions: sensory perception, moisture, activity, mobility, nutrition, and friction/shear. A total score of ≤12 indicates high risk of developing pressure injuries, 13-14 indicates moderate risk, and ≥15 indicates low risk.
Quality of life among older adults | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be assessed using the EQ-5D-5L questionnaire. The scale has two parts: a five-question survey and a visual analogue scale (VAS). The five questions measure health-related quality of life (HRQoL) in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) on a Likert scale (1 = no problems; 5 = extreme problems). Responses are converted into a single index value ranging from 0 (equivalent to death) to 1 (optimal health), applying Spanish population utility index values. The validated version for the general Spanish-speaking population will be used in this study.
Perceived social support | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be assessed using the DUKE-UNC-11 Perceived Social Support Questionnaire (DUKE-11). The DUKE-11 is self-administered and measures perceived functional social support across 11 items divided into two dimensions: 'confidential support' and 'affective support'. All items use a five-point Likert scale (1 = as much as desired; 5 = much less than desired) to indicate the frequency of social support received. Scores range from 11-55 points, with scores >32 indicating low perceived social support.
Loneliness | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Loneliness will be assessed using the three-item version of the UCLA Loneliness Scale (UCLA-3). The UCLA-3 measures subjective perception of loneliness through three items addressing key aspects of social disconnection. Participants respond using a three-point Likert scale (1 = never, 2 = sometimes, 3 = always). Total scores range from 3-9 points, with higher scores indicating greater perceived social isolation and lower scores indicating less loneliness.
Coping self-efficacy | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be assessed using the Coping Self-Efficacy Scale (CSES). This scale measures an individual's perceived confidence in their ability to manage stressful or challenging situations. It comprises 26 items, each rated on an 11-point Likert scale (0 = "cannot do at all," 10 = "can do without difficulty"), grouped into three dimensions: use of coping strategies, emotional control, and positive thinking. Higher scores indicate greater perceived self-efficacy in coping with stress.
Emotional status | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  This will be measured using the Hospital Anxiety and Depression Scale (HADS), which assesses levels of anxiety and depression. The scale consists of 14 questions with four response options (0-3 points), seven items relating to anxiety and seven to depression. The maximum score for each subscale is 21, with a total maximum of 42 points. Scores above 11 on each subscale indicate the presence of anxiety or depression.
Glycated hemoglobin (HbA1c) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  HbA1c (%) will be measured in blood samples as an indicator of long-term glucose metabolism.
Fasting blood glucose | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Fasting glucose concentration (mg/dL) will be measured in blood samples as an indicator of short-term glucose metabolism.
High-density lipoproteins (HDL) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum HDL cholesterol levels (mg/dL).
Low-density lipoproteins (LDL) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum LDL cholesterol levels (mg/dL).
Total cholesterol | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum total cholesterol levels (mg/dL).
Omega-3 polyunsaturated fatty acids (N-3 PUFA) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Plasma concentration of N-3 PUFA (µmol/L).
Serum albumin | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum albumin concentration (g/dL).
C-reactive protein (CRP) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum CRP concentration (mg/L).
Interleukin-6 (IL-6) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum IL-6 concentration (pg/mL)
Tumour necrosis factor-alpha (TNF-α) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum TNF-α concentration (pg/mL).
Gamma-glutamyl transferase (GGT) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum GGT activity (U/L).
Aspartate aminotransferase (AST) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum AST activity (U/L).
Alanine aminotransferase (ALT) | [Time Frame: T1=pre-test (immediately before being enrolled onto one of the groups); T2=post-test (between 1-12 days after the visit programme has been completed); T3=6-month follow-up (six months after finishing the intervention programme)]
  Serum ALT activity (U/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
A database with the participants' total scores for the study's primary and secondary outcome measures will be made available to other researchers once all the papers presenting the study's results have been published.
Supporting Information: Study Protocol
Time Frame: The study protocol will be made available to other researchers once it has been published in a scientific journal (estimated timeframe: starting December 2026) and will be available for 6 months.

REFERENCES:
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Lockwood EB, Schober M. Factors Influencing the impact of nurse practitioners' clinical autonomy: a self determining perspective. Int Nurs Rev. 2024 Jun;71(2):375-395. doi: 10.1111/inr.12948. Epub 2024 Apr 23. PMID 38651183
- [Background] Saunders R, Seaman K, Graham R, Christiansen A. The effect of volunteers' care and support on the health outcomes of older adults in acute care: A systematic scoping review. J Clin Nurs. 2019 Dec;28(23-24):4236-4249. doi: 10.1111/jocn.15041. Epub 2019 Sep 30. PMID 31429987
- [Background] de Sandes-Guimaraes LV, Dos Santos PC, Alves CPGP, Cervato CJ, Silva APA, Leao ER. The effect of volunteer-led activities on the quality of life of volunteers, residents, and employees of a long-term care institution: a cohort study. BMC Geriatr. 2023 Mar 20;23(1):151. doi: 10.1186/s12877-023-03898-y. PMID 36941534
- [Background] Jadczak AD, Makwana N, Luscombe-Marsh N, Visvanathan R, Schultz TJ. Effectiveness of exercise interventions on physical function in community-dwelling frail older people: an umbrella review of systematic reviews. JBI Database System Rev Implement Rep. 2018 Mar;16(3):752-775. doi: 10.11124/JBISRIR-2017-003551. PMID 29521871
- [Background] Garcia-Nogueras I, Aranda-Reneo I, Pena-Longobardo LM, Oliva-Moreno J, Abizanda P. Use of Health Resources and Healthcare Costs associated with Frailty: The FRADEA Study. J Nutr Health Aging. 2017;21(2):207-214. doi: 10.1007/s12603-016-0727-9. PMID 28112778
- [Background] Veronese N, Custodero C, Cella A, Demurtas J, Zora S, Maggi S, Barbagallo M, Sabba C, Ferrucci L, Pilotto A. Prevalence of multidimensional frailty and pre-frailty in older people in different settings: A systematic review and meta-analysis. Ageing Res Rev. 2021 Dec;72:101498. doi: 10.1016/j.arr.2021.101498. Epub 2021 Oct 23. PMID 34700009
- [Background] Rivas-Ruiz F, Machon M, Contreras-Fernandez E, Vrotsou K, Padilla-Ruiz M, Diez Ruiz AI, de Mesa Berenguer Y, Vergara I; Group GIFEA. Prevalence of frailty among community-dwelling elderly persons in Spain and factors associated with it. Eur J Gen Pract. 2019 Oct;25(4):190-196. doi: 10.1080/13814788.2019.1635113. Epub 2019 Oct 22. PMID 31637940
- [Background] Kojima G, Iliffe S, Walters K. Frailty index as a predictor of mortality: a systematic review and meta-analysis. Age Ageing. 2018 Mar 1;47(2):193-200. doi: 10.1093/ageing/afx162. PMID 29040347
- [Background] Gutierrez-Valencia M, Izquierdo M, Cesari M, Casas-Herrero A, Inzitari M, Martinez-Velilla N. The relationship between frailty and polypharmacy in older people: A systematic review. Br J Clin Pharmacol. 2018 Jul;84(7):1432-1444. doi: 10.1111/bcp.13590. Epub 2018 May 3. PMID 29575094
- [Background] Espinoza SE, Quiben M, Hazuda HP. Distinguishing Comorbidity, Disability, and Frailty. Curr Geriatr Rep. 2018 Dec;7(4):201-209. doi: 10.1007/s13670-018-0254-0. Epub 2018 Sep 19. PMID 30984516
- [Background] Milte R, Petersen J, Boylan J, Henwood T, Hunter S, Lange B, Lawless M, Torode S, Lewis LK. Prevalence and determinants of physical frailty among people living in residential aged care facilities: a large-scale retrospective audit. BMC Geriatr. 2022 May 14;22(1):424. doi: 10.1186/s12877-022-03101-8. PMID 35568811
- [Background] Kojima G. Frailty as a predictor of disabilities among community-dwelling older people: a systematic review and meta-analysis. Disabil Rehabil. 2017 Sep;39(19):1897-1908. doi: 10.1080/09638288.2016.1212282. Epub 2016 Aug 24. PMID 27558741
- [Background] Cesari M, Marzetti E, Thiem U, Perez-Zepeda MU, Abellan Van Kan G, Landi F, Petrovic M, Cherubini A, Bernabei R. The geriatric management of frailty as paradigm of "The end of the disease era". Eur J Intern Med. 2016 Jun;31:11-4. doi: 10.1016/j.ejim.2016.03.005. Epub 2016 Mar 18. PMID 26997416
- [Background] Holmberg C, Wolf A, Olsson MM, Heckemann B. Nurses' general attitudes and caregiving-specific perceptions toward the oldest-old: A nationwide survey. Int J Nurs Stud. 2022 Dec;136:104379. doi: 10.1016/j.ijnurstu.2022.104379. Epub 2022 Oct 10. PMID 36356546
- [Background] Hladek MD, Gill J, Bandeen-Roche K, Walston J, Allen J, Hinkle JL, Lorig K, Szanton SL. High coping self-efficacy associated with lower odds of pre-frailty/frailty in older adults with chronic disease. Aging Ment Health. 2020 Dec;24(12):1956-1962. doi: 10.1080/13607863.2019.1639136. Epub 2019 Jul 10. PMID 31290680
- [Background] Gale CR, Westbury L, Cooper C. Social isolation and loneliness as risk factors for the progression of frailty: the English Longitudinal Study of Ageing. Age Ageing. 2018 May 1;47(3):392-397. doi: 10.1093/ageing/afx188. PMID 29309502
- [Background] Cai Y, Han Z, Cheng H, Li H, Wang K, Chen J, Liu ZX, Xie Y, Lin Y, Zhou S, Wang S, Zhou X, Jin S. The impact of ageing mechanisms on musculoskeletal system diseases in the elderly. Front Immunol. 2024 May 7;15:1405621. doi: 10.3389/fimmu.2024.1405621. eCollection 2024. PMID 38774874
- [Background] Briones Peralta MÁ, Pardo García I, Escribano Sotos F. Políticas públicas de cuidados de larga duración: residencias para mayores, calidad del servicio y atención de calidad. Int Rev Econ Policy. 2021;3(1):76-98.
- [Background] Huesa Andrade M, Calvo-Gallego JL, Pedregal Gonzalez MA, Bohorquez Colombo P. [Differences between institutionalized patients and those included in a home care program in Seville]. Aten Primaria. 2020 Aug-Sep;52(7):488-495. doi: 10.1016/j.aprim.2019.10.002. Epub 2020 Feb 17. Spanish. PMID 32081457